CLINICAL TRIAL: NCT02546934
Title: A Phase III, Multicenter, Randomized Study of ABX Plus Cisplatin (AP) Versus Gemcitabine Plus Cisplatin (GP) as First-Line Treatment in Patients With Advanced Triple-Negative Breast Cancer
Brief Title: ABX Plus Cisplatin Versus Gemcitabine Plus Cisplatin in Triple Negative Breast Cancer (TNBC)
Acronym: TNBC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Dr, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2015-18 CBCSG018
Record Dates: First submitted 2015-09-10; First posted 2015-09-11 (Estimated); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: triple negative breast cancer; fine line chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABX, cisplatin (Experimental): AP (ABX and cisplatin combination)
  Interventions: Drug: ABX, cisplatin
- Gemcitabine, Cisplatin (Active Comparator): GP (Gemcitabine and Cisplatin combination)
  Interventions: Drug: Gemcitabine, Cisplatin

INTERVENTIONS:
Drug: ABX, cisplatin — ABX 125 mg/m2, IV drip 30 minutes, D1, D8 Cisplatin 75 mg/m2, IV drip 120 minutes, D1
  Other Names: experimental arm
  Arms: ABX, cisplatin
Drug: Gemcitabine, Cisplatin — Gemcitabine 1250 mg/m2, IV drip 30 minutes, D1, D8 Cisplatin 75 mg/m2, IV drip 120 minutes, D1
  Other Names: control arm
  Arms: Gemcitabine, Cisplatin

SUMMARY:
ABX Plus Cisplatin Versus Gemcitabine Plus Cisplatin in Triple Negative Breast Cancer (TNBC)

DETAILED DESCRIPTION:
A Phase III, Multicenter, Randomized Study of ABX Plus Cisplatin (AP) Versus Gemcitabine Plus Cisplatin (GP) as First-Line Treatment in Patients With Advanced Triple-Negative Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Females with age between 18 and 70 years old
2. Histological proven unresectable recurrent or advanced breast cancer, including de novo stage IV disease.
3. Triple-negative for estrogen receptor (ER), progestogen receptor (PR), and human epithelial receptor-2 (HER2) by immunohistochemistry (ER <1%, PR <1% and Her2 negative). A negative Her2 gene amplification should be verified by FISH test for those patients with Her2 (2+). For those with Her2 (1+), FISH test might be considered by the investigator.
4. No prior chemotherapy for metastatic breast cancer is permitted. Prior administration of chemotherapy in the adjuvant/neoadjuvant setting is acceptable if completed 6 months before the enrollment.
5. At least one measurable disease according to the response evaluation criteria in solid tumor (RECIST 1.1)
6. Performance status no more than 1
7. All patients enrolled are required to have adequate hematologic, hepatic, and renal function
8. Life expectancy longer than 12 weeks
9. No serious medical history of heart, lung, liver and kidney
10. Be able to understand the study procedures and sign informed consent.

Exclusion Criteria:

1. Pregnant or lactating women (female patients of child-bearing potential must have a negative serum pregnancy test within 14 days before the first day of drug dosing, or, if positive, a pregnancy should be ruled out by ultrasound)
2. Women of child-bearing potential, unwilling to use adequate contraceptive protection during the process of the study
3. Treatment with radiotherapy at the axial skeleton within 4 weeks before the first treatment or has not recovered from all toxicities of previous radiotherapy
4. Treatment with an investigational product within 4 weeks before the first treatment
5. Patients with symptomatic central nervous system metastases are not permitted, except for those with stable and asymptomatic brain metastases who have completed cranial irradiation, and have at least one measurable lesion outside the brain. Radiotherapy should be completed within 4 weeks prior to the registration
6. Other active malignancies (including other hematologic malignancies) or other malignancies within the last 5 years, except for cured nonmelanoma skin cancer or cervical intraepithelial neoplasia.
7. Patients having a history of clinically significant cardiovascular, hepatic, respiratory or renal diseases, clinically significant hematological and endocrinal abnormalities, clinically significant neurological or psychiatric conditions
8. Uncontrolled serious infection

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
PFS (Progression Free Survival) | 6 weeks

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 6 weeks
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 6 weeks
Overall Survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China

REFERENCES:
- [Derived] Wang B, Sun T, Zhao Y, Wang S, Zhang J, Wang Z, Teng YE, Cai L, Yan M, Wang X, Jiang Z, Pan Y, Luo J, Shao Z, Wu J, Guo X, Hu X. A randomized phase 3 trial of Gemcitabine or Nab-paclitaxel combined with cisPlatin as first-line treatment in patients with metastatic triple-negative breast cancer. Nat Commun. 2022 Jul 12;13(1):4025. doi: 10.1038/s41467-022-31704-7. PMID 35821019
- [Derived] Wang B, Zhao Y, Li Y, Xu Y, Chen Y, Jiang Q, Yao D, Zhang L, Hu X, Fu C, Zhang S, Chen S. A plasma SNORD33 signature predicts platinum benefit in metastatic triple-negative breast cancer patients. Mol Cancer. 2022 Jan 18;21(1):22. doi: 10.1186/s12943-022-01504-0. No abstract available. PMID 35042534